CLINICAL TRIAL: NCT00003856
Title: A Multicenter, Multi-National, Open-Label, Single Group, Single and Multiple Dose Study of Foscan-Mediated Photodynamic Therapy (PDT) for the Palliative Treatment of Recurrent, Refractory or Second Primary Squamous Cell Carcinomas of the Head and Neck in Patients Considered to be Incurable With Surgery or Radiotherapy
Brief Title: Photodynamic Therapy in Treating Patients With Recurrent, Refractory, or Second Primary Head and Neck Cancer That Cannot Be Treated With Surgery or Radiation Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Quintiles, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067019; QUINT-009.003.08b; SCOTIA-QUINT-009.003.08b; NCI-V99-1539
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-01

CONDITIONS: Head and Neck Cancer
Keywords: recurrent salivary gland cancer; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — temoporfin

INTERVENTIONS:
Drug: temoporfin

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. This may be an effective palliative treatment for head and neck cancer.

PURPOSE: Phase II trial to study the effectiveness of photodynamic therapy for palliative treatment in patients who have recurrent, refractory, or second primary head and neck cancer that cannot be treated with surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the individual clinical benefit of temoporfin-mediated photodynamic therapy for palliative treatment in patients with recurrent, refractory, or second primary squamous cell cancer of the head and neck. II. Determine the improvement in global, functional, and symptomatic measures of quality of life in these patients. III. Determine the toxic effects, tolerability, and safety of this regimen in these patients. IV. Determine the population pharmacokinetics, objective tumor response (complete and partial), and the 1 year survival of these patients on this regimen.

OUTLINE: This is a multicenter study. Patients receive IV temoporfin on day -4, followed by laser light therapy on day 0. Patients are treated every 4 to 16 weeks for a maximum of 3 courses. Patients are evaluated on days 1, 2, 7, and weeks 2, 4, 6, 8, 12, and 16 following laser light therapy. Quality of life is assessed at baseline through week 12 of follow-up. Patients are followed monthly for 4 months after the final treatment, then every 3 months for 1 year.

PROJECTED ACCRUAL: A minimum of 50 prospective and 25 retrospective patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent, refractory, or second primary squamous cell cancer of the head and neck that is incurable with surgery or radiotherapy Any N, Any M, single or multiple tumor(s) Locally accessible, discrete tumor(s) by CT or MRI scan Must be considered incurable with surgery or radiotherapy, for example: Distant disease (e.g., lung and/or liver metastases) OR Cervical disease fixed to surrounding structures (e.g., carotid artery or prevertebral fascia) OR Metastases in the site of prior radiotherapy OR Not suitable for anesthesia or reconstructive surgery OR Multiple cutaneous metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No disease exacerbated by light, including systemic lupus erythematosus, psoriasis, porphyria, actinic reticuloid, or xeroderma pigmentosum Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 30 days since prior chemotherapy (6 weeks since nitrosoureas) Endocrine therapy: Concurrent steroid therapy allowed Radiotherapy: At least 30 days since prior radiotherapy to the head and neck Surgery: At least 30 days since prior surgery and recovered Other: At least 30 days since prior light activated therapy or medication (e.g.,PUVA or Accutane) No prior photodynamic therapy At least 30 days since prior experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1998-10

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Larson, Study Chair — Quintiles, Inc.
Locations (7):
- United States (7):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Division of Head and Neck Surgery, Evanston, Illinois
  - Norton Healthcare Pavilion, Louisville, Kentucky
  - Ear, Nose, and Throat Specialty Care of Minnesota, P.A., Minneapolis, Minnesota
  - School of Dental Medicine, Buffalo, New York
  - St. Luke's-Roosevelt Hospital, New York, New York